CLINICAL TRIAL: NCT02621034
Title: Comparison of Post-endodontic Pain Using Reciproc and Oneshape Rotary Instrumentation Systems: A Randomized Clinical Trial
Brief Title: Comparative Evaluation of Post-endodontic Pain Using Two Rotary Instrumentation Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zahedan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SRH-1
Record Dates: First submitted 2015-11-29; First posted 2015-12-03 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-03

CONDITIONS: Pain
Keywords: Root canal treatment; pain; endodontic instruments
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Experimental): K-file hand instrumentation
  Interventions: Procedure: Control
- Reciproc (Experimental): rotary reciprocating protocol
  Interventions: Procedure: Reciproc
- One shape (Experimental): one shape continuous rotation protocol
  Interventions: Procedure: One shape

INTERVENTIONS:
Procedure: Control — K-file hand instrumentation
  Arms: Control
Procedure: Reciproc — reciprocating rotary instrument
  Arms: Reciproc
Procedure: One shape — full rotation protocol
  Arms: One shape

SUMMARY:
In this study the investigators aim to compare the post-operative pain using two single-file endodontic rotary systems : Reciproc and One shape.

DETAILED DESCRIPTION:
Comparison of the post operative pain with two rotary systems including Reciproc and One shape.

Confounding factors were neutralized and the rotary systems were compared.

ELIGIBILITY:
Inclusion Criteria:

* Systematically healthy patients
* First or second molars with irreversible pulpitis without periapical pathosis.
* Single visit endodontic treatment

Exclusion Criteria:

* Root canal retreatment
* Pregnancy
* The presence of a difficult root canal anatomy
* Internal or external resorption
* Teeth with open apices
* Any accident of complication occurred during treatment
* Presence of periapical lesion, abscess or sinus tract

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eshagh Ali Saberi, DDS,MS, Study Director — Head of the department of Endodontics, Zahedan university of medical sciences
Locations (1):
- Zahedan Dental School, Zahedan, Iran

RESULTS

PARTICIPANT FLOW:
Groups:
- k File: hand instrumentation
  k file: hand instrumentation
Period: Overall Study
Arm/Group | k File | Reciproc | One Shape
Started | 53 | 52 | 55
Completed | 50 | 50 | 50
Not Completed | 3 | 2 | 5
Not completed — Lost to Follow-up | 3 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Reciproc | One Shape | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (13.4) | 33.2 (13.7) | 30.2 (10.1) | 31.7 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 31 | 34 | 92
  Male | 23 | 19 | 16 | 58
Tooth type [Number; unit: participants]
  Maxillary molars | 25 | 11 | 20 | 56
  Mandibular molars | 25 | 39 | 30 | 94

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain on the Visual Anlogue Scale (VAS) at the 6-hour Post-operative Interval
Description: The pain VAS is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10).
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Reciproc | One Shape
Number analyzed (Participants) | 50 | 50 | 50
units on a scale | 5 (2.8) | 3.2 (3.1) | 3.5 (2.9)

2. Primary Outcome: Comparison of Post-operative Pain in the Reciproc and Oneshape Groups Through Out the Intervals
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reciproc | One Shape
Number analyzed (Participants) | 50 | 50
units on a scale | 0.46 (0.26) | 0.34 (0.15)

3. Primary Outcome: Comparison of Post-operative Pain Between the Three Groups at the 72-hour Interval
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Reciproc | One Shape
Number analyzed (Participants) | 50 | 50 | 50
units on a scale | 0.72 (0.19) | 0.46 (0.26) | 0.34 (0.15)

ADVERSE EVENTS:
Description: Serious and Other [Not Including Serious] Adverse Events were not collected/assessed.
Arm/Group | Control | Reciproc | One Shape
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No